CLINICAL TRIAL: NCT05083312
Title: An Adolescent Sub-study Within FLUTE-2: A Randomized, Double-blind, Placebo-Controlled Study of APT-1011 (Fluticasone Propionate Oral Dispersible Tablet Formulation), With an Open-label Extension, in Adolescent Subjects With Eosinophilic Esophagitis
Brief Title: Efficacy and Safety APT-1011 in Adolescent Subjects With Eosinophilic Esophagitis (EoE) - A Sub-Study of the FLUTE-2 Trial
Acronym: FLUTEEN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ellodi Pharmaceuticals, LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SP-1011-003a
Record Dates: First submitted 2021-10-06; First posted 2021-10-19 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Eosinophilic Esophagitis
Keywords: APT-1011; Esophagitis; Eosinophilic Esophagitis; Esophageal Diseases; Gastrointestinal Diseases; Gastroenteritis; Eosinophilia; Leukocyte Disorders; Hematologic Diseases; Hypersensitivity, Immediate; Hypersensitivity; Immune System Diseases; Fluticasone; Anti-Inflammatory Agents; Bronchodilator Agents; Autonomic Agents; Peripheral Nervous System Agents; Anti-Asthmatic Agents; Respiratory System Agents; Anti-Allergic Agents
MeSH Terms: conditions — Eosinophilic Esophagitis; Esophagitis; Esophageal Diseases; Gastrointestinal Diseases; Gastroenteritis; Eosinophilia; Leukocyte Disorders; Hematologic Diseases; Hypersensitivity, Immediate; Hypersensitivity; Immune System Diseases | interventions — APT-1011; Fluticasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- APT-1011 (Experimental): APT-1011 3 mg HS
  Interventions: Drug: APT-1011
- Placebo (Placebo Comparator): HS
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: APT-1011 — APT-1011 is an orally disintegrating tablet that includes fluticasone propionate as its active ingredient.
  Other Names: fluticasone propionate
  Arms: APT-1011
Drug: Placebo oral tablet — Placebo orally disintegrating tablet
  Other Names: PBO
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled study of APT-1011, followed by an open-label extension (OLE) in adolescents (≥12 to <18 years) with EoE.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled study of APT-1011, followed by an open-label extension (OLE) in adolescents (≥12 to <18 years) with EoE that will evaluate the efficacy and safety of APT-1011 3 mg administered HS for the induction of response to treatment (histologic and symptomatic) over 12 weeks.

At Week 12, subjects may move into the open-label single arm study of APT-1011 3 mg hora somni (HS; at bedtime). All subjects who do not move into the open-label study will return at Week 14 for a 2-week off-treatment follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥12 and <18 years of age
2. Each subject and their parents or legal guardian, must read, understand and provide consent or assent on the ICF for this study and be willing and able to adhere to study-related treatment regimens, procedures and visit schedule
3. Diagnosis or presumptive diagnosis of EoE that is confirmed during the Screening period by histology that demonstrates ≥15 peak eos/HPF. In order to ensure that a diagnosis can be made, at least 6 biopsies should be taken from both proximal and distal specimens (at least 3 each). Mid-esophageal biopsies are not required (optional). HPF will be defined as a standard area of 235 square microns in a microscope with 40x lens [0.3 mm^2] and 22 mm ocular.

   1. Esophagogastroduodenoscopies and biopsies are to be obtained during the Screening period
   2. Biopsies will be read by a central pathologist
   3. Esophagogastroduodenoscopies and biopsies performed outside the study will not be accepted to meet eligibility criteria
   4. Optional biopsies may be taken and processed locally for local use, only where specified in the local ICF. If serious pathology is unexpectedly encountered, biopsies of such lesions must be processed locally
4. Have a subject-reported history of ≥6 episodes of dysphagia in the 14 days prior to baseline
5. Completion of the daily diary on at least 11 out of the 14 days during the 2-week Baseline Symptom Assessment

Exclusion Criteria:

1. Have known contraindication, hypersensitivity, or intolerance to corticosteroids
2. Have a contraindication to, or factors that substantially increase the risk of, EGD procedure or esophageal biopsy or have narrowing of the esophagus that precludes EGD with a standard 9 mm endoscope at screening
3. Have history of an esophageal stricture requiring dilatation within the 12 weeks prior to Screening
4. Bone mineral density >2 SD below height-adjusted for age
5. Have any physical, mental, or social condition or history of illness or laboratory abnormality that in the Investigator's judgment might interfere with study procedures or the ability of the subject to adhere to and complete the study or increase the safety risk to the subject such as uncontrolled diabetes or hypertension or may increase risk of corticosteroid toxicity (e.g., abnormal bone mineral density)
6. History of recurrent (persistent) or current oral or esophageal mucosal infection due to inhaled or nasal corticosteroids
7. Have any mouth or dental condition that prevents normal eating (excluding braces)
8. Have any condition affecting the esophageal mucosa or altering esophageal motility other than EoE, including erosive esophagitis (grade B or higher as per the Los Angeles Classification of Gastroesophageal Reflux Disease, hiatus hernia longer than 3 cm, Barrett's esophagus, and achalasia)
9. Use of systemic (oral or parenteral) corticosteroids within 60 days before Screening, use of swallowed corticosteroids within 30 days before Screening
10. Initiation of either inhaled or nasal corticosteroids or high-potency dermal topical corticosteroids within 30 days before Screening
11. Use of calcineurin inhibitors or purine analogues (azathioprine, 6-mercaptopurine) in the 12 weeks before Screening
12. Use of potent CYP 3A4 inhibitors (e.g., ritonavir and ketoconazole) in the 12 weeks before Screening
13. Initiation of an elimination diet or elemental diet within 30 days before Screening (diet must remain stable after signing ICF)
14. Morning (07:00 to 09:00, or as close to that window as possible) serum cortisol level ≤5 μg/dL (138 nmol/L) that is not responsive to ACTH stimulation: defined as a serum cortisol level <16 μg/dL (440 nmol/L) at 60 minutes with ACTH stimulation test using 250 μg cosyntropin (i.e., an abnormal result on the ACTH stimulation test)
15. Use of biologic immunomodulators in the 24 weeks before Screening (environmental allergen desensitization injection or oral therapy (excluding food allergen desensitization) is allowed as long as the course of therapy is not altered during the study period)
16. Subjects who have initiated, discontinued, or changed dosage regimen of histamine H2 receptor antagonists, antacids or antihistamines, leukotriene inhibitors or sodium cromolyn within 4 weeks before qualifying endoscopy during Screening. If already receiving these drugs, the dosage must remain constant throughout the study
17. Subjects who have changed dosage regimen of PPIs within 8 weeks before qualifying endoscopy. If already receiving PPIs, the dosage must remain constant throughout the study
18. Infection with hepatitis B, hepatitis C, or human immunodeficiency virus
19. Have gastrointestinal bleeding or documented active peptic ulcer within 4 weeks prior to Screening or entering a new study period
20. Have chronic infection such as prior or active tuberculosis, active chicken pox or measles or absence of prior measles, mumps and rubella vaccine. Subjects with tuberculosis exposure or who live in, or travel to, high endemic areas should be assessed locally for tuberculosis before consideration for the study
21. Immunosuppression or immunodeficiency disorder
22. Current malignancy or malignancy within 3 years of Screening. Subjects in remission for at least 3 years post-treatment may be enrolled.
23. Known severe bleeding disorder
24. Have a history or presence of Crohn's disease, celiac disease, or other inflammatory disease of the gastrointestinal tract, including eosinophilic gastroenteritis
25. Have current drug abuse in the opinion of the Investigator.
26. Have current alcohol abuse in the opinion of the Investigator.
27. Female subjects who are pregnant, breastfeeding, or planning to become pregnant during the study
28. Sexually active females of childbearing potential who do not agree to follow highly effective contraceptive methods through the End of Study visit
29. Have received an investigational product, as part of a clinical trial within 30 days (or 5 half-lives, whichever is longest) of Screening. Subjects who are currently participating in observational studies or enrolled in patient registries are allowed in this study
30. Have participated in a prior study with investigational product APT-1011

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2021-09-30 (Actual); Primary Completion 2022-09-05 (Actual); Study Completion 2022-09-05 (Actual)

PRIMARY OUTCOMES:
Week 12 histologic responder rates | Week 12
  To compare the Week 12 histologic responder rates (≤ 6 peak eosinophils / high power field [eos/HPF]) for APT-1011 3 mg hora somni (HS) with that for placebo. HPF will be defined as a standard area of 235 square microns in a microscope with 40x lens [0.3 mm^2] and 22 mm ocular
Mean change in number of dysphagia episodes | Week 0 to Week 12
  To compare the mean change in number of dysphagia episodes from baseline to Week 12 for APT-1011 3 mg HS with that for placebo

SECONDARY OUTCOMES:
Mean change in EREFs from Week 0 to Week 12 | Week 0 to Week 12
  To compare endoscopic appearance evaluated by the mean change from baseline to Week 12 in Eosinophilic Esophagitis Endoscopic Reference Score (EREFs) for APT-1011 3 mg HS with that for placebo. The EREF score has a range from 0-9, with 9 being worst result.
Percentage of subjects with <1 peak eos/HPF at Week 12 | Week 12
  To compare the percentage of subjects with <1 peak eos/HPF at Week 12 for APT-1011 3 mg HS with that for placebo
Mean change in PROSE Symptom Burden Score | Week 0 to Week 12
  To compare the mean change from baseline to Week 12 in the day-level symptom burden using the Patient Reported Outcomes Symptoms of EoE (PROSE) for APT-1011 3 mg HS with that for placebo
Mean change in PROSE day-level difficulty swallowing | Week 0 to Week 12
  To compare the mean change from baseline to Week 12 in day-level difficulty swallowing using the PROSE for APT-1011 3 mg HS with that for placebo
Histologic Change from Baseline to Week 12 | Week 0 to Week 12
  To compare mean histologic change from baseline to Week 12 for APT-1011 3 mg HS with that for placebo
Percentage of subjects with <15 peak eos/HPF | Week 12
  To compare the percentage of subjects with <15 peak eos/HPF at Week 12 for APT-1011 3 mg HS with that for placebo
Mean number of dysphagia-free days | Week 0 to Week 12
  To compare the mean number of dysphagia-free days from baseline to Week 12 for APT-1011 3 mg HS with that for placebo

CONTACTS AND LOCATIONS:
Overall Officials: Mirna Chehade, MD, MPH, Principal Investigator — Mount Sinai Center for Eosinophilic Disorders
Locations (3):
- United States (2):
  - IU School of Medicine Department of Pediatrics, Indianapolis, Indiana
  - Boston Specialists, Boston, Massachusetts
- Royal Children's Hospital, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No